CLINICAL TRIAL: NCT00427154
Title: Effect of Inhaled Pre-Prandial Human Insulin Plus Metformin & Glimepiride Versus Rosiglitazone Plus Metformin & Glimepiride on HbA1c in Subjects With Type 2 Diabetes
Brief Title: Effect of Inhaled Pre-prandial Human Insulin on Blood Glucose Control in Type 2 Diabetes
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: See termination reason in detailed description
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN1998-1540
Record Dates: First submitted 2007-01-25; First posted 2007-01-26 (Estimated); Last update posted 2018-09-05 (Actual); Status verified 2018-09

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Rosiglitazone; Metformin; glimepiride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator)
  Interventions: Drug: inhaled human insulin; Drug: metformin; Drug: glimepiride
- B (Active Comparator)
  Interventions: Drug: rosiglitazone; Drug: metformin; Drug: glimepiride

INTERVENTIONS:
Drug: rosiglitazone — Tablets, 4 mg once or twice daily.
  Arms: B
Drug: inhaled human insulin — Treat-to-target dose titration scheme, inhalation.
  Other Names: NN1998
  Arms: A
Drug: metformin — Tablets, 2000 mg/day.
Drug: glimepiride — Tablets, 8 mg/day.

SUMMARY:
This trial is conducted in the United States of America (USA). This trial will compare the changes in HbA1c after 26 weeks of inhaled insulin or rosiglitazone treatment, both in combination with metformin and glimepiride.

DETAILED DESCRIPTION:
The decision to discontinue the development of AERx® is not due to any safety concerns. An analysis concluded that fast-acting inhaled insulin in the form it is known today, is unlikely to offer significant clinical or convenience benefits over injections of modern insulin with pen devices.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* Currently treated with antidiabetes drugs (including Exenatide) for at least 2 months
* HbA1c between 7.5 and 11.0% (both inclusive) on antidiabetes combination therapy
* BMI less than or equal to 40 kg/m2

Exclusion Criteria:

* Current smoking or smoking within the last 6 months
* Current acute or chronic pulmonary disease (except for asthma)
* Proliferative retinopathy requiring acute treatment
* Clinically significant disease history including kidney or liver disease
* Heart disease which limits physical activity or results in discomfort with physical activity
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 227 (Actual)
Dates: Start 2007-01-10 (Actual); Primary Completion 2008-03-11 (Actual); Study Completion 2008-03-11 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c | After 26 weeks

SECONDARY OUTCOMES:
Fasting plasma glucose | For the duration of the trial
Lipid profiles | For the duration of the trial
Hypoglycaemic episodes | For the duration of the trial
Glucose profiles | For the duration of the trial
Change in body weight | For the duration of the trial

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (98):
- United States (98):
  - Novo Nordisk Investigational Site, Hueytown, Alabama
  - Novo Nordisk Investigational Site, Ozark, Alabama
  - Novo Nordisk Investigational Site, Tuscaloosa, Alabama
  - Novo Nordisk Investigational Site, Vestavia Hills, Alabama
  - Novo Nordisk Investigational Site, Tucson, Arizona
  - Novo Nordisk Investigational Site, Concord, California
  - Novo Nordisk Investigational Site, Escondido, California
  - Novo Nordisk Investigational Site, Fresno, California
  - Novo Nordisk Investigational Site, Huntington Beach, California
  - Novo Nordisk Investigational Site, La Jolla, California
  - Novo Nordisk Investigational Site, Orange, California
  - Novo Nordisk Investigational Site, Poway, California
  - Novo Nordisk Investigational Site, Roseville, California
  - Novo Nordisk Investigational Site, Sacramento, California
  - Novo Nordisk Investigational Site, San Diego, California
  - Novo Nordisk Investigational Site, Santa Barbara, California
  - Novo Nordisk Investigational Site, Temecula, California
  - Novo Nordisk Investigational Site, Walnut Creek, California
  - Novo Nordisk Investigational Site, Colorado Springs, Colorado
  - Novo Nordisk Investigational Site, Waterbury, Connecticut
  - Novo Nordisk Investigational Site, Boca Raton, Florida
  - Novo Nordisk Investigational Site, Clearwater, Florida
  - Novo Nordisk Investigational Site, Hialeah, Florida
  - Novo Nordisk Investigational Site, Hollywood, Florida
  - Novo Nordisk Investigational Site, Lake Mary, Florida
  - Novo Nordisk Investigational Site, Marianna, Florida
  - Novo Nordisk Investigational Site, Melbourne, Florida
  - Novo Nordisk Investigational Site, Merritt Island, Florida
  - Novo Nordisk Investigational Site, Miami, Florida
  - Novo Nordisk Investigational Site, Palm Harbor, Florida
  - Novo Nordisk Investigational Site, Pembroke Pines, Florida
  - Novo Nordisk Investigational Site, Vero Beach, Florida
  - Novo Nordisk Investigational Site, West Palm Beach, Florida
  - Novo Nordisk Investigational Site, Athens, Georgia
  - Novo Nordisk Investigational Site, Atlanta, Georgia
  - Novo Nordisk Investigational Site, Augusta, Georgia
  - Novo Nordisk Investigational Site, Dunwoody, Georgia
  - Novo Nordisk Investigational Site, Powder Springs, Georgia
  - Novo Nordisk Investigational Site, Roswell, Georgia
  - Novo Nordisk Investigational Site, Suwanee, Georgia
  - Novo Nordisk Investigational Site, Tucker, Georgia
  - Novo Nordisk Investigational Site, Honolulu, Hawaii
  - Novo Nordisk Investigational Site, Boise, Idaho
  - Novo Nordisk Investigational Site, Chicago, Illinois
  - Novo Nordisk Investigational Site, Peoria, Illinois
  - Novo Nordisk Investigational Site, Springfield, Illinois
  - Novo Nordisk Investigational Site, Lafayette, Indiana
  - Novo Nordisk Investigational Site, Des Moines, Iowa
  - Novo Nordisk Investigational Site, Shawnee Mission, Kansas
  - Novo Nordisk Investigational Site, Topeka, Kansas
  - Novo Nordisk Investigational Site, Wichita, Kansas
  - Novo Nordisk Investigational Site, Lexington, Kentucky
  - Novo Nordisk Investigational Site, Scarborough, Maine
  - Novo Nordisk Investigational Site, Baltimore, Maryland
  - Novo Nordisk Investigational Site, Marlborough, Massachusetts
  - Novo Nordisk Investigational Site, Springfield, Massachusetts
  - Novo Nordisk Investigational Site, Jackson, Mississippi
  - Novo Nordisk Investigational Site, Chesterfield, Missouri
  - Novo Nordisk Investigational Site, Jefferson City, Missouri
  - Novo Nordisk Investigational Site, Kansas City, Missouri
  - Novo Nordisk Investigational Site, St Louis, Missouri
  - Novo Nordisk Investigational Site, Billings, Montana
  - Novo Nordisk Investigational Site, Omaha, Nebraska
  - Novo Nordisk Investigational Site, Las Vegas, Nevada
  - Novo Nordisk Investigational Site, Berlin, New Jersey
  - Novo Nordisk Investigational Site, Cherry Hill, New Jersey
  - Novo Nordisk Investigational Site, Lawrenceville, New Jersey
  - Novo Nordisk Investigational Site, Staten Island, New York
  - Novo Nordisk Investigational Site, Syracuse, New York
  - Novo Nordisk Investigational Site, Asheville, North Carolina
  - Novo Nordisk Investigational Site, Charlotte, North Carolina
  - Novo Nordisk Investigational Site, Greenville, North Carolina
  - Novo Nordisk Investigational Site, High Point, North Carolina
  - Novo Nordisk Investigational Site, Cincinnati, Ohio
  - Novo Nordisk Investigational Site, Cleveland, Ohio
  - Novo Nordisk Investigational Site, Dayton, Ohio
  - Novo Nordisk Investigational Site, Clinton, Oklahoma
  - Novo Nordisk Investigational Site, Oklahoma City, Oklahoma
  - Novo Nordisk Investigational Site, Medford, Oregon
  - Novo Nordisk Investigational Site, Altoona, Pennsylvania
  - Novo Nordisk Investigational Site, Beaver, Pennsylvania
  - Novo Nordisk Investigational Site, Norristown, Pennsylvania
  - Novo Nordisk Investigational Site, Greer, South Carolina
  - Novo Nordisk Investigational Site, Chattanooga, Tennessee
  - Novo Nordisk Investigational Site, Clarksville, Tennessee
  - Novo Nordisk Investigational Site, Kingsport, Tennessee
  - Novo Nordisk Investigational Site, Arlington, Texas
  - Novo Nordisk Investigational Site, Dallas, Texas
  - Novo Nordisk Investigational Site, Houston, Texas
  - Novo Nordisk Investigational Site, Hurst, Texas
  - Novo Nordisk Investigational Site, Lewisville, Texas
  - Novo Nordisk Investigational Site, San Antonio, Texas
  - Novo Nordisk Investigational Site, Arlington, Virginia
  - Novo Nordisk Investigational Site, Norfolk, Virginia
  - Novo Nordisk Investigational Site, Richmond, Virginia
  - Novo Nordisk Investigational Site, Warrenton, Virginia
  - Novo Nordisk Investigational Site, Renton, Washington
  - Novo Nordisk Investigational Site, Tacoma, Washington

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com